CLINICAL TRIAL: NCT05538260
Title: Epidemiology and Visual Outcome of Pediatric Ocular Trauma
Brief Title: Pediatric Ocular Trauma in Minia Governate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hosny Ahmed Zein, DR, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MiniaU PED
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Ocular Trauma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Repair of ocular trauma in children below 16 years old — Diagnosis and repair of pediatric ocular trauma

SUMMARY:
The most common cause of unilateral blindness in pediatric age groups, especially in developing countries, is ocular trauma. The epidemiology of eye injuries varies in different parts of the world and different age groups and depends on many factors including life style, socioeconomic status, traffic state, sport and creative activities and type of registration and recording of data. About half a million people in the world are blind as a result of eye injuries. About 30-40% of monocular blindness is due to ocular trauma

ELIGIBILITY:
Inclusion Criteria:

* Age below 16 years

Exclusion Criteria:

* Age above 16 years Previous ocular surgery

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of trauma | 2 years
  incidence of trauma
Visual outcome | 6 months
  Visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No